CLINICAL TRIAL: NCT05571046
Title: Efficacy of Intramuscular Glucocorticoid Injection in Patients With Lumbar Radicular Pain
Brief Title: Glucocorticoid Injection in Patients With Lumbar Radicular Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Sibel Basaran, Head of Physical Medicine and Rehabilitation, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cukurova14980; TTU-2022-14980 (Other Grant/Funding Number: Cukurova University)
Record Dates: First submitted 2022-09-30; First posted 2022-10-07 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Radiculopathy Lumbar
Keywords: glucocorticoid; radicular pain; lumbar radiculopathy
MeSH Terms: conditions — Radiculopathy | interventions — Glucocorticoids; betamethasone dipropionate, betamethasone sodium phosphate drug combination

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glucocorticoid injection (Active Comparator): Intramuscular glucocorticoid (5 mg betamethasone dipropionate and 2 mg betamethasone sodium phosphate)
  Interventions: Drug: Glucocorticoids
- Placebo injection (Placebo Comparator): Intramuscular saline (%0.9 isotonic sodium chloride)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Glucocorticoids — Intramuscular injection of single dose of 1 ml betamethasone, Paracetamol (500 mg, 2 times a day)
  Other Names: Diprospan
  Arms: Glucocorticoid injection
Other: Placebo — Intramuscular injection of %0.9 isotonic sodium chloride, Paracetamol (500 mg, 2 times a day)
  Arms: Placebo injection

SUMMARY:
The purpose of this study is to demonstrate the efficacy of intramuscular betamethasone injection on pain and other clinical parameters in patients with radicular pain due to lumbar disc herniation. The investigators also aimed to determine the effects on electrophysiological findings.

DETAILED DESCRIPTION:
Low back pain is an important health problem that causes difficulties in daily living activities, loss of work performance and disability. Some patients with low back pain have radicular symptoms due to intervertebral disc herniation. Lumbar radiculopathy is characterized by radiating buttock and leg pain in a lumbar nerve root distribution.

The pathophysiology of radiculopathy is related to compression of the nerve, as well as the local release of inflammatory cytokines. Systemic corticosteroids have been used for treatment of lumbar radicular pain for a long time. The effects of corticosteroids are related to their anti-inflammatory effects, which may help reduce swelling and related compression on the affected nerve. Corticosteroids can be used systemically (i.e. oral, intravenous, or intramuscular routes) or administered directly into spinal structures through injections.

In the current study, the investigators aimed to demonstrate the efficacy of intramuscular betamethasone injection on pain, disability and health related quality of life in patients with lumbar radicular pain due to disc herniation. The investigators also aimed to determine the effects on electrophysiological findings.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 65 years old with acute (less than 6 weeks) lumbar radicular pain due to intervertebral disc herniation.
* Neurological findings such as sensory, motor and reflex abnormality matching the L4, L5 or S1 nerve distribution.
* Patients who confirmed to have root compression (radiculopathy) by electrophysiological investigations.

Exclusion Criteria:

* Contraindication for steroid usage (acute infection, uncontrolled diabetes and hypertension, severe cardiac failure), hypersensitivity to steroids
* Acute trauma
* Inflammatory low back pain
* Indications for neurosurgery (pronounced motor weakness or cauda equina syndrome)
* Lumbar spinal stenosis
* History of back surgery, history of steroid injection in the last 3 months
* Pregnancy, lactation
* Malignancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2023-10-26 (Actual)

PRIMARY OUTCOMES:
Lumbar radicular pain | Week 1
  Visual analog scale (VAS, min-max values: 0-100, higher scores mean a worse outcome)
Lumbar radicular pain | Month 1
  Visual analog
  (VAS, min-max values: 0-100, higher scores mean a worse outcome)
Lumbar radicular pain | Month 3
  Visual analog
  (VAS, min-max values: 0-100, higher scores mean a worse outcome)
Disability | Month 1
  Oswestry Disability Index
  (ODI, min-max values: 0-100, higher scores mean a worse outcome)
Disability | Month 3
  Oswestry Disability Index
  (ODI, min-max values: 0-100, higher scores mean a worse outcome)
Health related quality of Life | Month 1
  Nottingham Health Profile
  (NHP, 6 subscales, for each subscale min-max values: 0-100, higher scores mean a worse outcome)
Health related quality of Life | Month 3
  Nottingham Health Profile (NHP, 6 subscales, for each subscale min-max values: 0-100, higher scores mean a worse outcome)

SECONDARY OUTCOMES:
Electrophysiological evaluation (Sensory NCS) | Month 1
  Sensory nerve conduction study (m/s)
Electrophysiological evaluation (Motor NCS) | Month 1
  Motor nerve conduction study (m/s)
Electrophysiological evaluation (F wave) | Month 1
  F wave (m/s)
Electrophysiological evaluation (H reflex) | Month 1
  H reflex (m/s)

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Basaran, MD, Prof, Study Director — Cukurova University
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

REFERENCES:
- [Derived] Boga Vijdan E, Basaran S, Balal M. Efficacy of intramuscular glucocorticoid injection in patients with lumbar radicular pain: a randomized controlled trial. BMC Musculoskelet Disord. 2025 Jul 4;26(1):650. doi: 10.1186/s12891-025-08897-1. PMID 40616084